CLINICAL TRIAL: NCT02468778
Title: Supporting Patients Undergoing HIgh-Risk PCI Using a High-Flow PErcutaneous Left Ventricular Support Device (SHIELD II)
Brief Title: SHIELD II Clinical Investigation
Acronym: SHIELD II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Abbott has decided to discontinue our percutaneous heart pump (PHP) program and the SHIELD II trial because the product was not meeting the needs of the patients it was intended to serve.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10148 Ver. J
Record Dates: First submitted 2015-05-29; First posted 2015-06-11 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease
Keywords: HeartMate PHP; High Risk PCI; Mechanical circulatory support device; MCS; Abbott; SJM-CIP-10148
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- HeartMate PHP (Roll-in) (Experimental): Participants who receive a HeartMate PHP device without randomisation will be included in this arm
  Interventions: Device: HeartMate PHP
- HeartMate PHP (Randomised) (Experimental): Participants who receive a HeartMate PHP device after randomisation will be included in this arm
  Interventions: Device: HeartMate PHP
- Any Abiomed Impella® (Randomised) (Active Comparator): Participants who receive any Abiomed Impella® Device approved for use in high-risk PCI after randomisation will be included in this arm
  Interventions: Device: Any Abiomed Impella® device approved for use in high-risk PCI

INTERVENTIONS:
Device: HeartMate PHP — The HeartMate PHP System is a temporary (<6 hours) ventricular assist device indicated for use during high-risk percutaneous coronary interventions (PCI) performed electively or urgently in hemodynamically stable patients with severe coronary artery disease, when a heart team, including a cardiac surgeon, has determined high-risk PCI is an acceptable therapeutic option. Use of the HeartMate PHP Systems in these patients may prevent hemodynamic instability, which can result from repeat episodes of reversible myocardial ischemia that occur during planned temporary coronary occlusions and may reduce peri-and post-procedural adverse events.
  Arms: HeartMate PHP (Randomised); HeartMate PHP (Roll-in)
Device: Any Abiomed Impella® device approved for use in high-risk PCI — Any Abiomed Impella® device approved for use in high-risk PCI.
  Arms: Any Abiomed Impella® (Randomised)

SUMMARY:
The HeartMate PHP System is a temporary (<6 hours) ventricular assist device indicated for use during high-risk percutaneous coronary interventions (PCI) performed electively or urgently in hemodynamically stable patients with severe coronary artery disease, when a heart team, including a cardiac surgeon, has determined high-risk PCI is the appropriate therapeutic option. Use of the HeartMate PHP Systems in these patients may prevent hemodynamic instability, which can result from repeat episodes of reversible myocardial ischemia that occur during planned temporary coronary occlusions and may reduce peri-and post-procedural adverse events.

DETAILED DESCRIPTION:
Prospective, randomized, multi-center, open-label trial of the HeartMate PHP at up to 120 sites in the United States (U.S.). Control device will be any Abiomed Impella device approved for use in high-risk PCI.

This clinical investigation is divided into two phases, a feasibility phase and a pivotal phase.

* Feasibility Phase: Includes 75 roll-in and 120 randomized subjects registered under the clinical investigational plan (CIP) versions 2-4 at 48 sites in the U.S. prior to January 30, 2017
* Pivotal Phase: Includes subjects to be registered under Version F or a later version of the CIP at up to 120 sites in the U.S.

Non-randomized Roll-in Cohort: Up to 480 subjects with the HeartMate PHP.

Randomized Cohort: A minimum of 473 and a maximum of 716 subjects will be randomized in a 2:1 ratio to the HeartMate PHP and Impella.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Subject is undergoing elective or urgent high-risk PCI procedure and is hemodynamically stable
* Subject is indicated for a revascularization of at least one de novo or restenotic lesion in a native coronary vessel or bypass graft
* A heart team, including a cardiac surgeon, has determined high risk PCI is an acceptable therapeutic option
* Subject must provide written informed consent prior to any clinical investigation related procedure

Imaging Inclusion Criteria:

• The presence of complex coronary artery disease (CAD) makes hemodynamic instability resulting from repeat episodes of reversible myocardial ischemia during PCI likely. Complex CAD is defined as an ejection fraction of <50% by echocardiographic assessment AND at least one of the following:

* intervention of the last patent coronary conduit, OR
* intervention of an unprotected left main artery, OR
* intervention on patient presenting with triple vessel disease defined as at least one significant stenosis (at least 50% diameter stenosis on visual assessment) in all three major epicardial territories

Exclusion Criteria:

* Emergency PCI
* Any prior coronary revascularization within the last 6 months
* Any MI with elevated cardiac biomarker (creatinine kinase-MB (CK-MB) or troponin >1X upper limit of normal (ULN)) and no evidence of at least 1 consecutive CK-MB or troponin value trending downward from previous value (at least 4 hours apart) OR ST Elevation MI (STEMI) within 72 hours prior to the index procedure regardless of the level of cardiac biomarker
* Cardiac arrest within 24 hours of procedure requiring cardiopulmonary resuscitation (CPR) or defibrillation
* Any use of a mechanical circulatory support device within 14 days prior to the index procedure (Note: Subjects must be hemodynamically stable without any hemodynamic support to be eligible for this clinical investigation.)
* Hemodynamic support with a mechanical circulatory support device (e.g.,the HeartMate PHP, Impella, intra-aortic balloon pump (IABP), or extracorporeal membrane oxygenation (ECMO)), post-PCI is anticipated
* Any condition that requires discontinuation of antiplatelet and/or anticoagulant therapy within 90 days following the index procedure (e.g., planned noncardiac surgery)
* Any use of vasopressors or inotropes within 24 hours prior to the index procedure
* Staged PCI is planned within 90 days following device removal
* Cardiogenic shock (SBP <90 mmHg for >1 hour with either cool clammy skin OR oliguria OR altered sensorium AND cardiac index <2.2 L/min/m^2)
* History of aortic valve replacement or repair
* Severe peripheral vascular disease that will preclude the use of a 14F access sheath, which is required for the insertion of the HeartMate PHP catheter (If the investigator is unsure of the presence or severity of the peripheral vascular diseases for study device access, an appropriate imaging assessment (e.g., duplex ultrasound, angiogram or computerized tomography) should be performed to verify the access before randomization.)
* Known abnormalities of the aorta that would preclude surgery, including aneurysms and significant tortuosity or calcifications
* Subject is on hemodialysis
* Liver dysfunction with elevation of liver enzymes and bilirubin levels to ≥ 3X ULN or Internationalized Normalized Ratio (INR) ≥1.6 or lactate dehydrogenase (LDH) > 2.5X ULN
* Abnormal coagulation parameters (platelet count ≤75000/mm^3 or INR ≥1.6 or fibrinogen ≤1.5 g/l)
* Active systemic infection requiring treatment with antibiotics
* Subject had active COVID-19 symptoms and/or a positive test result within the prior 2 months
* Stroke or transient ischemic attack (TIA) within 6 months of procedure
* Any allergy or intolerance to ionic and nonionic contrast media, anticoagulants (including heparin), or antiplatelet therapy drugs that cannot be adequately premedicated
* Subject is pregnant (For a female subject of childbearing potential, a pregnancy test must be performed within 14 days (≤14 days) prior to the index procedure per site standard test)
* Participation in another clinical study of an investigational drug or device that has not met its primary endpoint
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with followup requirements, or impact the scientific soundness of the clinical investigation results
* Life expectancy <1 year

Imaging Exclusion Criteria:

* Mural thrombus in the left ventricle
* Documented presence of aortic stenosis (orifice area of 1.5 cm^2 or less)
* Moderate to severe aortic insufficiency by echocardiographic assessment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Coe, Study Director — Abbott
Locations (58):
- United States (58):
  - Scottsdale Shea Medical Center, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - USC University Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - St.Joseph Hospital, Orange, California
  - University of Miami, Miami, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Iowa Heart Center, West Des Moines, Iowa
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Mercy Medical Research Institute, Springfield, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Maimonides, Brooklyn, New York
  - New York University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Medical Center Clinical Sciences, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Seton Medical Center, Austin, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 PHP roll-in and 36 randomized subjects were registered at 15 sites in the pivotal phase of the study.
Period: Overall Study
Arm/Group | HeartMate PHP (Roll-in) | HeartMate PHP (Randomised) | Any Abiomed Impella® (Randomised)
Started | 18 | 26 | 10
Completed | 15 | 22 | 7
Not Completed | 3 | 4 | 3
Not completed — Death | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HeartMate PHP (Roll-in) | HeartMate PHP (Randomised) | Any Abiomed Impella® (Randomised) | Total
Number analyzed (Participants) | 18 | 26 | 10 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (8.7) | 67.8 (8.8) | 72.2 (6.7) | 70.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 2 | 10
  Male | 15 | 21 | 8 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 1 | 8
  Not Hispanic or Latino | 15 | 14 | 6 | 35
  Unknown or Not Reported | 1 | 7 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 1 | 4 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 0 | 1 | 4
  White | 12 | 17 | 4 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 26 | 10 | 54
Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 12 | 11 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participants With Composite of Cardiovascular Death, Myocardial Infarction, Stroke, Any Unplanned Repeat Revascularization (PCI/CABG), Bleeding (BARC 3/5) up to 14 Days Post-device Removal, Severe Hypotension, and Change in Aortic Insufficiency
Description: The primary endpoint, including the following components representing important safety and effectiveness endpoints will be evaluated using the difference in event rates in the ITT population.
  * Cardiovascular Death
  * Myocardial infarction (MI)
  * Stroke
  * Any unplanned repeat revascularization (PCI or CABG)
  * Bleeding (BARC 3 or 5) up to 14 days post-device removal
  * Severe hypotension, defined as: systolic blood pressure (SBP) or augmented diastolic pressure (whichever is greater) <90 mmHg while on device support requiring (1) more than one administration of OR (2) continuous infusion of inotropic/pressor medications to restore hemodynamics
  * Change in aortic insufficiency from baseline to 90 days by echocardiographic assessment.
Time Frame: 90 Days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percentage of participants
Arm/Group | HeartMate PHP (Roll-in) | HeartMate PHP (Randomised) | Any Abiomed Impella® (Randomised)
Number analyzed (Participants) | 17 | 21 | 4
percentage of participants | 29.4 | 19.0 | 50.0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | HeartMate PHP (Roll-in) | HeartMate PHP (Randomised) | Any Abiomed Impella® (Randomised)
All-Cause Mortality (participants affected / at risk) | 2/18 | 1/26 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/18 | 9/26 | 5/10
Other Adverse Events (participants affected / at risk) | 8/18 | 8/26 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HeartMate PHP (Roll-in) (N=18) | HeartMate PHP (Randomised) (N=26) | Any Abiomed Impella® (Randomised) (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Thrombosis (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 2 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Arthritis Infective (Infections and infestations) | 0 | 1 | 0
Corona Virus Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 2 | 0 | 1
Troponin Increased (Investigations) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 2 | 0
Shock Haemorrhagic (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HeartMate PHP (Roll-in) (N=18) | HeartMate PHP (Randomised) (N=26) | Any Abiomed Impella® (Randomised) (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Corona Virus Infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision Site Hemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 2 | 1 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 2 | 0
Cardiac Enzymes Increased (Investigations) | 4 | 8 | 3
Free Hemoglobin Present (Investigations) | 1 | 2 | 0
Hemoglobin Decreased (Investigations) | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 1 | 0
Troponin Increased (Investigations) | 1 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Major Depression (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arterial Occlusive Disease (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0
Haemorrhage (Vascular disorders) | 2 | 1 | 0
Hypotension (Vascular disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish or present results of its performance of the Study consistent with the terms of this section. If the Study is part of a multi-center clinical study, Institution agrees that the first publication of results will be made as a joint multi-center publication with investigators from all sites contributing data.

DOCUMENTS (2):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02468778/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02468778/SAP_001.pdf